CLINICAL TRIAL: NCT03098654
Title: Impact of Integrated HIV/NCD Screening on HIV Testing Uptake and Engagement in HIV Care: an RCT in Kisarawe, Tanzania
Brief Title: Impact of Integrated HIV/NCD Screening on HIV Testing Uptake and Engagement in HIV Care in Kisarawe, Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00064733; 1R01MH111366-01 (NIH)
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Human Immunodeficiency Virus; Diabetes Mellitus, Type 2; Hypertension
Keywords: Human Immunodeficiency Virus; Community Health Services; Chronic Disease; Integrated Delivery of Health Care; Tanzania
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Diabetes Mellitus, Type 2; Hypertension; Chronic Disease | interventions — Diet; Health Services Needs and Demand; Metformin; Thiazides

STUDY DESIGN:
Intervention Model Description: Once two similar HIV Care and Treatment Centers (CTCs) are matched, they will be randomized to receive either the intervention or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Intervention (Experimental): Members will have DM and HTN managed at the CTC together with their HIV care. Interventions include:
  1. Community mobilization activities to inform community members of available services
  2. Support at the local health center to aid clinicians in managing uncontrolled cases of DM and HTN, including training for clinical staff, glucometers/test strips, and BP monitors.
  3. HIV counseling and serial rapid HIV testing
  4. Blood glucose and blood pressure testing
  5. DM/HTN medications as needed
  6. Personalized diet and lifestyle counseling for all participants with elevated glucose or BP that includes education, dietary assessment and recommendations, advice on physical activity, and the need to regularly monitor their glucose/BP.
  Interventions: Diagnostic Test: Blood glucose and blood pressure testing; Behavioral: Diet and lifestyle counseling; Drug: DM/HTN medications as needed
- Control (No Intervention): Members in the control arm will receive community-level rapid HIV testing at the CTCs, which is the standard of care. HIV testing performed by the CTC is according to the National HIV Testing Algorithm (serial rapid testing using Determine HIV 1/2 and Uni-Gold HIV 1/2) which follows Tanzanian and international (WHO/CDC) standards for provision of HIV counseling and testing. Those who test positive for HIV will be referred to the CTC for the standard Tanzanian level of HIV care, which includes counseling and ART medication managed at the CTCs.

INTERVENTIONS:
Diagnostic Test: Blood glucose and blood pressure testing — Diabetes will be assessed using a 6-question risk assessment on a 10-point scale (based on a field-tested and culturally adapted International Diabetes Federation formula on DM risk factors and symptoms) and a random blood glucose test with a portable finger stick glucose monitor. Those with either: (1) a risk score of 5 or more, or (2) a random blood glucose with a value greater than 140 mg/dl, will be asked to return after fasting for at least 8 hours to have a fasting glucose test taken. Blood pressure will be assessed using a portable battery operated automatic BP cuff. The BP test will include three values taken at least 5-minutes apart and the 3 will be averaged to determine the final value.
  Other Names: Biosense V2 monitor; Lifesource 767 PV
  Arms: Enhanced Intervention
Behavioral: Diet and lifestyle counseling — All participants with elevated glucose or BP will receive personalized lifestyle counseling by trained counselors informed by lab results and that includes education on diabetes, hypertension, dietary assessment and recommendations, advice on physical activity, and the need to regularly monitor their glucose, BP, and adjust their diet, activity level, as needed. Personalized risk reduction plans will be negotiated with the client during their scheduled visits.
  Arms: Enhanced Intervention
Drug: DM/HTN medications as needed — Subjects will receive DM or HTN medications prescribed by the CTC clinician as needed.
  Other Names: Glucophage; Metformin; Thiazide
  Arms: Enhanced Intervention

SUMMARY:
This study focuses on the integration of HIV and NCD screening and care. The investigators will conduct a randomized controlled trial examining the efficacy and cost-effectiveness of the intervention strategy in Kisarawe District, Tanzania, a rural area 40 KM southwest of Dar es Salaam. The study will match two similar HIV care and treatment centers (CTC) in the District, one of which will be randomized to receive the enhanced intervention which will integrate diabetes (DM) and hypertension (HTN) screening with the existing HIV testing program, and integrate care for DM and HTN into the HIV care program. Comparisons of the community HIV testing rates in the two communities, engagement in HIV care among those testing positive, and 24-month retention in HIV care will be assessed among a cohort of 107 newly enrolled patients per community.

Specifically, the aims are to determine:

1. Whether integrating DM and HTN screening with HIV testing will increase the uptake of community-level HIV testing.
2. If integrating DM/HTN care with HIV care enhances engagement in HIV care.
3. Whether integration of DM/HTN care with HIV care enhances retention in HIV care for those newly enrolled in HIV care.
4. The cost-effectiveness of integrating NCD screening and care with HIV screening and care with regard to the incremental cost per HIV infected client engaged in HIV care, and cost per newly enrolled HIV client retained in HIV care over 24-months.

ELIGIBILITY:
Eligibility Criteria for Screening:

• Be aged 18 years or above.

Inclusion Criteria for Intervention and Control Cohorts:

* Be aged 18 years or above.
* Recently enrolled in HIV care and treatment

Exclusion Criteria:

* Potentially vulnerable populations (incarcerated, under age of consent, unable to understand the procedures planned, etc.).
* Individuals under the influence of drugs or alcohol and anyone presenting with mental disability that would preclude ability to understand study procedure, risks, and benefits.
* Inability or unwillingness of subject to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Uptake of community-level HIV testing | 12 months
  Uptake of HIV testing will be measured as the annual cumulative number of unique persons receiving HIV testing as a proportion of the community size in each HIV CTC venue using clinic records from the government CTC.
Engagement in HIV care | 12 months
  Engagement will be measured as proportion of persons testing positive for HIV who advance to successful enrollment in HIV care at the CTC. Persons will be documented with biometric fingerprint matching against those who tested for HIV in the study area. Comparisons will be made across the enhanced and comparison CTCs.
Retention in HIV care | 24 months
  Retention in HIV care will be measured in several ways, including the Human Resources and Services Administration HIV/AIDS Bureau definition of 2 or more outpatient visits at least 3-months apart during each year, the number of missed clinic visits, and appointment adherence (number of completed visits/number of scheduled visits) during the study period.

SECONDARY OUTCOMES:
Adherence to DM/HTN/ARV medication | 24 months
  Self-reported medication adherence questions adapted from our other NIH-funded study (Dyadic-Based Diagnosis, Care, and Prevention for HIV Discordant Couples) will be used to assess medication adherence. The Self-Reported Medication Nonadherence Measurement tool will be used to assess reasons for nonadherence.
Adherence to physical activity intervention | 24 months
  Global Physical Activity Questionnaire (GPAQ) to assess DM / HTN lifestyle changes for NCD positive subjects in the intervention arm. The GPAQ is a 12-item survey created by the World Health Organization to measure physical activity (intensity, duration, and frequency) and domains of performance (related to occupation, transportation, and leisure).
Adherence to dietary intervention | 24 months
  A food frequency questionnaire developed for use specifically in Tanzania and surrounding countries will be used to assess dietary changes.
Biological, Psychological, and Social adverse events associated with the study intervention | 24 months
  Self-reported and staff-reported adverse events (biological, psychological, or social) experienced as an outcome of receiving the intervention.
Cost-effectiveness of integrating NCD screening and care with HIV screening and care | 24 months
  Cost will be measured through regular cost worksheets that the investigators will collect throughout the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Sweat, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No